CLINICAL TRIAL: NCT04839354
Title: Sickle Cell Disease Treatment With Arginine Therapy (STArT) Trial
Acronym: STArT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Claudia R. Morris (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Claudia R. Morris, Professor, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00002344; PECARN Protocol Number 050 (Other: Pediatric Emergency Care Applied Research Network); UG3HL148560 (NIH)
Record Dates: First submitted 2021-04-08; First posted 2021-04-09 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Sickle Cell Disease
Keywords: Arginine Therapy; Pain management
MeSH Terms: conditions — Anemia, Sickle Cell; Agnosia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-Arginine Hydrochloride (Experimental): Participants receiving L-arginine hydrochloride in parenteral form. Participants receive up to 21 doses, with participants who are discharged early receiving fewer doses.
  Interventions: Drug: L-Arginine Hydrochloride
- Placebo (Placebo Comparator): Participants receiving normal saline as a placebo for L-arginine hydrochloride for up to 21 doses, with participants who are discharged early receiving fewer doses.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: L-Arginine Hydrochloride — A one-time L-arginine hydrochloride loading dose of 200 mg/kg will be administered intravenously (IV) followed by a standard dose of 100 mg/kg given by IV three times per day (TID).
  Arms: L-Arginine Hydrochloride
Other: Normal saline — A placebo of normal saline will be administered by IV with a loading dose of 2ml/kg followed by 1ml/kg given by IV three times per day (TID).
  Arms: Placebo

SUMMARY:
The trial is designed to test intravenous (IV) arginine therapy in children with sickle cell disease (SCD) and vaso-occlusive painful episodes (VOE) to further knowledge on efficacy and safety of this orphan drug.

DETAILED DESCRIPTION:
Pain is a clinical hallmark of sickle cell disease (SCD), and a significant problem in emergency medicine. Vaso-occlusive painful episodes (VOE) are common, debilitating, and a medical emergency. VOE are the leading cause of hospitalizations, emergency department (ED) visits, missed school, and are associated with an increased mortality rate. Symptomatic relief with analgesics and hydration are the only currently available treatments, and these have not changed in decades. Episodic periods of severe pain lead to high use of health care resources, with high readmission rates. A 2010 health care utilization report revealed that 20% of patients with SCD experienced ≥3 ED encounters per year. Hospital admission rates for VOE are approximately 60% for children with SCD and VOE. Many children with SCD also live with daily pain to some extent that their families try to control at home through various methods. It is when the pain becomes acutely worse, and unbearable, that they present to the ED in acute distress.

A significant evidence gap exists for best treatment of VOE and novel approaches to SCD/VOE that can be utilized in the ED and hospital ward are critically needed. Interventions that target underlying mechanisms of SCD pain in addition to providing symptomatic relief are worth pursuing.

Vaso-occlusion is believed to be the root cause of sickle cell pain. Nitric oxide (NO) is a free radical and a potent vasodilator that regulates vascular homeostasis and plays a role in SCD vaso-occlusion. NO has properties that can impact every aspect of SCD, and NO dysregulation is a common denominator among varied mechanisms of sickle vasculopathy. NO is produced in the endothelium from its obligate substrate L-arginine, which is converted to citrulline by a family of enzymes, the NO synthases (NOS). Although NOS expression and activity is increased, SCD is characterized by a state of NO resistance, NO inactivation, and impaired NO bioavailability. Under conditions of increased hemolysis, inflammation or oxidative stress, the compensatory upregulation of NO likely becomes overwhelmed and ineffective. Vascular dysfunction is the end result, due to complex and multifactorial interactions.

SCD is an arginine deficiency syndrome. Normal arginine metabolism is impaired for many reasons. Plasma arginine concentration decreases significantly in both adults and children with VOE and is associated with low nitric oxide (NO) and nitrogen dioxide (NO2) levels (NOx). It was observed that lowest arginine levels were found in children requiring admission for VOE, with arginine levels returning to baseline during convalescence in the hospital. Of interest, low plasma arginine concentration alone was a sensitive predictor for admission, while NOx levels were not, suggesting a function for arginine bioavailability in VOE severity that goes beyond NO. Although adults with SCD are arginine deficient at steady-state, children have plasma levels that are similar to normal controls. Alterations in the arginine metabolome differ in children vs. adults. An arginine deficiency develops with age and is influenced by acute events and chronic end organ damage that worsens over time. Children may therefore be more responsive to arginine therapy during an acute pain event compared to adults.

Arginine is a safe nutritional supplement that is FDA approved in parenteral form for growth hormone stimulation testing, with nearly 50 years of safety experience through its common use by endocrinologists. Experience with both oral and parenteral arginine therapy in sickle cell disease is growing. When arginine is given to SCD patients at steady-state, a paradoxical decrease in NOx occurs that is not overcome by higher doses, clearly indicating that arginine is metabolized differently in SCD compared to controls. However when arginine is given during VOE, a robust dose-dependent increase in NOx is observed. This indicates that arginine is also metabolized differently in SCD at steady-state (baseline) compared to times of acute illness including pain. Low dose arginine therapy is likely to be subtherapeutic in SCD; higher levels of plasma arginine are likely needed to overcome multi-factorial effects on global arginine bioavailability, and accelerated arginine consumption during VOE compared to baseline.

The trial is designed as a double-blind, placebo controlled, randomized, phase 3, multi-center trial of IV arginine therapy in children with VOE in SCD to further knowledge on efficacy and safety of the therapy. The exploratory objective is to more fully characterize the arginine metabolome in children with SCD during VOE, and evaluate the effects of arginine therapy on global arginine bioavailability and mitochondrial function together with important clinical outcomes of time to VOE resolution, pain scores, total parenteral opioid use, Patient-Reported Outcomes (PROs), and hospital length of stay in children with SCD and VOE.

Participants are randomized to receive 21 doses of IV arginine or a placebo, administered over 7 to 8 days (depending on what time of day the study drug was first administered on Day 1). Participants will be followed for up to 28 days following hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3-21 years of age, inclusive
2. Established diagnosis of sickle cell disease (any genotype)
3. Pain requiring medical care in an acute care setting (emergency department, hospital ward, day hospital, clinic) not attributable to non-sickle cell causes, treated with parenteral opioids

Exclusion Criteria:

1. Responds to 2 doses of IV opioids sufficiently for outpatient management
2. Greater than 12 hours from first dose of intravenous opioids to treat current pain in acute care setting
3. Hemoglobin less than 5 gm/dL or emergent need for red blood cell transfusion for hemodynamically unstable patient
4. Ketamine use in the emergency department for treatment of VOE
5. Glutamine within 30 days
6. New SCD drug use < 3 months (e.g. Hydroxyurea, voxelotor, crizanlizumab, etc)
7. Acute mental status or neurological changes
8. Acute stroke or clinical concern for stroke
9. Three or more ED visits for sickle cell related pain receiving parenteral opioids in previous 7 days (not including current emergency department visit)
10. Hospital discharge within previous 7 days
11. Hypotension requiring clinical intervention; hemodynamic instability; septic shock
12. Previous randomization in this arginine phase 3 randomized controlled trial
13. Use of inhaled nitric oxide, sildenafil or arginine within the last month
14. Non-English speaking or requires a translator for clinical care
15. Pregnancy
16. Allergy to arginine
17. PI/clinical team concerns for compliance/issues that may adversely impact study participation/outcome
18. Adults 18 years or older who lack medical decision-making capacity to consent

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 271 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Morris, MD, Principal Investigator — Emory University
Locations (10):
- United States (10):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta at Hughes Spalding, Atlanta, Georgia
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Washington University/St. Louis Children's Hospital, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital/Baylor College of Medicine, Houston, Texas
  - Medical College of Wisconsin/Wisconsin Children's Hospital, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results published for this study will be made available for sharing with other researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual participant data will be made available for sharing after publication of findings from this study
Access Criteria: Interested investigators can request de-identified data by sending an email to the principal investigator.

REFERENCES:
- [Background] Korman R, Hatabah D, Brown LA, Harris F, Wilkinson H, Rees CA, Bakshi N, Archer DR, Dampier C, Morris CR. Impact of arginine therapy on kyotorphin in children with sickle cell disease and vaso-occlusive pain. Blood Adv. 2024 Jun 25;8(12):3267-3271. doi: 10.1182/bloodadvances.2023012209. PMID 38527291
- [Background] Onalo R, Cilliers A, Cooper P, Morris CR. Arginine Therapy and Cardiopulmonary Hemodynamics in Hospitalized Children with Sickle Cell Anemia: A Prospective, Double-blinded, Randomized Placebo-controlled Clinical Trial. Am J Respir Crit Care Med. 2022 Jul 1;206(1):70-80. doi: 10.1164/rccm.202108-1930OC. PMID 35426778
- [Background] Reyes LZ, Figueroa J, Leake D, Khemani K, Kumari P, Bakshi N, Lane PA, Dampier C, Morris CR. Safety of intravenous arginine therapy in children with sickle cell disease hospitalized for vaso-occlusive pain: A randomized placebo-controlled trial in progress. Am J Hematol. 2022 Jan 1;97(1):E21-E24. doi: 10.1002/ajh.26396. Epub 2021 Nov 12. No abstract available. PMID 34724240
- [Background] Morris CR, Brown LAS, Reynolds M, Dampier CD, Lane PA, Watt A, Kumari P, Harris F, Manoranjithan S, Mendis RD, Figueroa J, Shiva S. Impact of arginine therapy on mitochondrial function in children with sickle cell disease during vaso-occlusive pain. Blood. 2020 Sep 17;136(12):1402-1406. doi: 10.1182/blood.2019003672. PMID 32384147
- [Background] Onalo R, Cooper P, Cilliers A, Vorster BC, Uche NA, Oluseyi OO, Onalo VD, Zubairu Y, Ayodele-Kehinde AU, Damilare OM, Figueroa J, Morris CR. Randomized control trial of oral arginine therapy for children with sickle cell anemia hospitalized for pain in Nigeria. Am J Hematol. 2021 Jan;96(1):89-97. doi: 10.1002/ajh.26028. Epub 2020 Nov 20. PMID 33075179
- [Background] Morris CR, Kato GJ, Poljakovic M, Wang X, Blackwelder WC, Sachdev V, Hazen SL, Vichinsky EP, Morris SM Jr, Gladwin MT. Dysregulated arginine metabolism, hemolysis-associated pulmonary hypertension, and mortality in sickle cell disease. JAMA. 2005 Jul 6;294(1):81-90. doi: 10.1001/jama.294.1.81. PMID 15998894
- [Background] Morris CR, Kuypers FA, Lavrisha L, Ansari M, Sweeters N, Stewart M, Gildengorin G, Neumayr L, Vichinsky EP. A randomized, placebo-controlled trial of arginine therapy for the treatment of children with sickle cell disease hospitalized with vaso-occlusive pain episodes. Haematologica. 2013 Sep;98(9):1375-82. doi: 10.3324/haematol.2013.086637. Epub 2013 May 3. PMID 23645695
- [Background] Sadeghi A, Taherifard E, Dehdari Ebrahimi N, Rafiei E, Hadianfard F, Taherifard E. Effects of l-arginine supplementation in patients with sickle cell disease: A systematic review and meta-analysis of clinical trials. Health Sci Rep. 2023 Apr 11;6(4):e1167. doi: 10.1002/hsr2.1167. eCollection 2023 Apr. PMID 37064309
- [Background] Onalo R, Cilliers A, Cooper P. Impact of oral L-arginine supplementation on blood pressure dynamics in children with severe sickle cell vaso-occlusive crisis. Am J Cardiovasc Dis. 2021 Feb 15;11(1):136-147. eCollection 2021. PMID 33815929
- [Background] Morris CR, Morris SM Jr, Hagar W, Van Warmerdam J, Claster S, Kepka-Lenhart D, Machado L, Kuypers FA, Vichinsky EP. Arginine therapy: a new treatment for pulmonary hypertension in sickle cell disease? Am J Respir Crit Care Med. 2003 Jul 1;168(1):63-9. doi: 10.1164/rccm.200208-967OC. Epub 2003 Mar 5. PMID 12626350
- [Result] Rees CA, Brousseau DC, Cohen DM, Villella A, Dampier C, Brown K, Campbell A, Chumpitazi CE, Airewele G, Chang T, Denton C, Ellison A, Thompson A, Ahmad F, Bakshi N, Coleman KD, Leibovich S, Leake D, Hatabah D, Wilkinson H, Robinson M, Casper TC, Vichinsky E, Morris CR; SCD Arginine Study Group and PECARN. Sickle Cell Disease Treatment with Arginine Therapy (STArT): study protocol for a phase 3 randomized controlled trial. Trials. 2023 Aug 17;24(1):538. doi: 10.1186/s13063-023-07538-z. PMID 37587492
- [Derived] Bolarinwa AB, Oduwole O, Okebe J, Ogbenna AA, Otokiti OE, Olatinwo AT. Antioxidant supplementation for sickle cell disease. Cochrane Database Syst Rev. 2024 May 22;5(5):CD013590. doi: 10.1002/14651858.CD013590.pub2. PMID 38775255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ten children's hospitals in the United States. Participant enrollment began June 21, 2021 and all follow-up assessments were completed by July 11, 2024.
Groups:
- L-Arginine Hydrochloride: Participants receiving L-arginine hydrochloride in parenteral form. Participants receive up to 21 doses, with participants who are discharged early receiving fewer doses. A one-time L-arginine hydrochloride loading dose of 200 mg/kg is administered intravenously (IV) followed by a standard dose of 100 mg/kg given by IV three times per day (TID).
- Placebo: Participants receiving normal saline as a placebo for L-arginine hydrochloride for up to 21 doses, with participants who are discharged early receiving fewer doses. A placebo of normal saline is administered by IV with a loading dose of 2ml/kg followed by 1ml/kg given by IV three times per day (TID).
Period: Overall Study
Arm/Group | L-Arginine Hydrochloride | Placebo
Started | 129 | 142
Completed | 129 | 142
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | L-Arginine Hydrochloride | Placebo | Total
Number analyzed (Participants) | 129 | 142 | 271
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14.8 [11.6 to 18.1] | 15.2 [10.7 to 17.7] | 15.1 [11.2 to 17.7]
Age, Customized [Count of Participants; unit: Participants]
  Under 12 years old | 36 | 42 | 78
  12 to 21 years old | 93 | 100 | 193
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 62 | 132
  Male | 59 | 80 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 7 | 20
  Not Hispanic or Latino | 115 | 135 | 250
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 115 | 134 | 249
  White | 3 | 5 | 8
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 7 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 129 | 142 | 271

OUTCOME MEASURES:

1. Primary Outcome: Time-to-crisis Resolution
Description: The time-to-crisis resolution is defined as the time in hours from the date and time of the first study drug delivery to time of the last dose of parenteral opioid delivery.
Time Frame: From study drug delivery to last IV opioid treatment (up to 1,724.1 hours)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | L-Arginine Hydrochloride | Placebo
Number analyzed (Participants) | 129 | 142
hours | 81.5 (79.6) | 88.6 (152.2)

2. Secondary Outcome: Total Parenteral Opioid Use
Description: Total parenteral opioid use is assessed as morphine equivalents in milligrams per kilogram (mg/kg).
Time Frame: From the time of IV placement throughout opioid treatment (up to 1,724.1 hours)
Measure: Mean (Standard Deviation); unit: milligrams per kilogram (mg/kg)
Arm/Group | L-Arginine Hydrochloride | Placebo
Number analyzed (Participants) | 129 | 142
milligrams per kilogram (mg/kg) | 2.6 (4.5) | 1.9 (2.8)

3. Secondary Outcome: Change in Pain Score
Description: Pain is assessed using a scale from 0 to 10, where 10 is the highest pain level. Daily highest and lowest pain scores are recorded. The change in score is calculated by subtracting the score at discharge from the score at the time of presentation.
Time Frame: Time of presentation and on the day of discharge (up to 554.8 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | L-Arginine Hydrochloride | Placebo
Number analyzed (Participants) | 129 | 142
score on a scale | 3.5 (3.3) | 3.7 (3.3)

4. Secondary Outcome: Change in Patient-Reported Outcome Measurement Information System (PROMIS) Pain Interference Score
Description: The PROMIS Pain Interference instrument is an 8-item, self-administered survey that assesses the interference of pain on daily activities. Participants are asked to respond to questions regarding the extent of their pain. Responses range from 1 to 5, where 1 represents "not at all" and 5 represents "very much". Total raw scores are converted to T-scores. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Scores below 50 indicate a lower amount of pain interference compared to the reference population, while scores higher than 50 indicate greater pain interference compared to the reference population. The change in score is calculated by subtracting the score at the time of discharge from the score from within 12 hours of study drug delivery. The change in score is calculated by subtracting the score at discharge from the score within 12 hours of study drug delivery.
Time Frame: Within 12 hours of study drug delivery, and on the day of discharge (up to 554.8 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | L-Arginine Hydrochloride | Placebo
Number analyzed (Participants) | 129 | 142
score on a scale | 3.5 (3.3) | 3.7 (3.3)

5. Secondary Outcome: Change in PROMIS Pain Behavior Score
Description: The PROMIS Pain Behavior instrument is an 8-item, self-administered survey that assesses external manifestations of pain. Participants are asked to respond to questions regarding the extent of their pain. Responses range from 1 to 5, where 1 represents "never" and 5 represents "always". Total raw scores are converted to T-scores. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Scores below 50 indicate a lower amount of pain behavior compared to the reference population, while scores higher than 50 indicate greater pain behavior compared to the reference population. The change in score is calculated by subtracting the score at discharge from the score within 12 hours of study drug delivery.
Time Frame: Within 12 hours of study drug delivery, and on the day of discharge (up to 554.8 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | L-Arginine Hydrochloride | Placebo
Number analyzed (Participants) | 129 | 142
score on a scale | 0.8 (6.8) | 1.0 (7.1)

6. Secondary Outcome: Change in PROMIS Fatigue Score
Description: The PROMIS Fatigue instrument is an 8-item, self-administered survey that assesses fatigue level within the past seven days. Participants are asked to respond to questions regarding fatigue frequency. Responses range from 1 to 5, where 1 represents "never" and five represents "always". Total raw scores are converted to T-scores. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Scores below 50 indicate a lower amount of fatigue compared to the reference population, while scores higher than 50 indicate greater fatigue compared to the reference population. The change in score is calculated by subtracting the score at discharge from the score within 12 hours of study drug delivery.
Time Frame: Within 12 hours of study drug delivery and on the day of discharge (up to 554.8 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | L-Arginine Hydrochloride | Placebo
Number analyzed (Participants) | 129 | 142
score on a scale | -0.4 (8.1) | 0.1 (9.1)

7. Other Pre Specified Outcome: Medication Quantification Score (MQS)
Description: Medication Quantification Score (MQS) is a tool to objectively quantify pain. The MQS is a validated score calculated based off of daily doses of pain related medications (including acetaminophen, aspirin, NSAIDs, and antidepressants). The MQS is a single numeric value for a patient's pain medication profile. This number is used to track pain levels through a treatment course.
Time Frame: Pre-dose and on day of discharge (up to 2 months)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Hospital Length of Stay
Description: Hospital length of stay in days is recorded.
Time Frame: Up to 6 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Pediatric PROMIS Score
Description: The Pediatric PROMIS assesses five domains of health with in a 35-item instrument. The survey is completed by patients ages 8-17 years of age and parents of children ages 5-17 years of age. The domains included are: pain behavior (8 items), pain interference (8 items), pain intensity (1 item), physical stress experiences (8 items), and fatigue (10 items). Total raw scores are converted to T-scores. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Scores below 50 indicate a lower amount of the concept being measured compared to the reference population, while scores higher than 50 indicate a greater amount of the concept being measured (e.g., more fatigue) compared to the reference population.
Time Frame: Within 12 hours of study drug delivery and on the day of discharge (up to 2 months)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: PedsQL SCD Pain and Hurt Scale Score
Description: The Pain and Hurt scale of the PedsQL SCD module has 9 items asking how much of a problem each item has been during the past month. Responses to items are given on a 5-point Likert scale where 0 = never a problem and 4 = almost always a problem. Items are reversed and transformed to a scale of 0 to 100 then the mean score for the scale is calculated. The total score for the Pain and Hurt scale ranges from 0 to 100 with higher scores indicating greater quality of life and lower SCD symptoms.
Time Frame: Within 12 hours of study drug delivery and on the day of discharge (up to 2 months)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: PedsQL SCD Pain Impact Scale Score
Description: The Pain Impact scale of the PedsQL SCD module has 10 items asking how much of a problem each item has been during the past month. Responses to items are given on a 5-point Likert scale where 0 = never a problem and 4 = almost always a problem. Items are reversed and transformed to a scale of 0 to 100 then the mean score for the scale is calculated. The total score for the Pain Impact scale ranges from 0 to 100 with higher scores indicating greater quality of life and lower SCD symptoms.
Time Frame: Within 12 hours of study drug delivery and on the day of discharge (up to 2 months)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Arginine Bioavailability
Description: Peak plasma arginine concentration is assessed via pharmacokinetic study.
Time Frame: Pre-Dose, Day 2, after 21 doses (Day 7 or 8) or at discharge (if discharged prior to Dose 21)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Mitochondrial Function
Description: Mitochondrial respiratory complex activities are measured to estimate mitochondrial function.
Time Frame: Pre-Dose, Day 2, after 21 doses (Day 7 or 8) or at discharge (if discharged prior to Dose 21)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time of randomization through Day 9 or hospital discharge or emergency department discharge (whichever comes first, up to 9 days). Emergency department revisits and hospital admissions were tracked through 28 days following hospital or emergency discharge and entered as adverse events or serious adverse events (up to 583 days).
Arm/Group | L-Arginine Hydrochloride | Placebo
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/142
Serious Adverse Events (participants affected / at risk) | 22/129 | 25/142
Other Adverse Events (participants affected / at risk) | 81/129 | 83/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | L-Arginine Hydrochloride (N=129) | Placebo (N=142)
Pain (General disorders) | 6 | 9
Sickle cell anaemia with crisis (General disorders) | 10 | 8
Acidosis (Blood and lymphatic system disorders) | 1 | 0
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Drug dependence (General disorders) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 1
Hallucination (General disorders) | 0 | 1
Intensive care (General disorders) | 1 | 0
Intentional overdose (Psychiatric disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | L-Arginine Hydrochloride (N=129) | Placebo (N=142)
Abdomial pain (General disorders) | 10 | 5
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Decreased appetite (General disorders) | 10 | 5
Decreased haemoglobin (Blood and lymphatic system disorders) | 12 | 5
Headache (General disorders) | 15 | 14
Hypoxemia (Blood and lymphatic system disorders) | 7 | 11
Nausea (General disorders) | 23 | 23
Pyrexia (General disorders) | 18 | 18
Vomiting (Gastrointestinal disorders) | 10 | 14
Transfusion (Blood and lymphatic system disorders) | 10 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT04839354/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT04839354/ICF_000.pdf